CLINICAL TRIAL: NCT05837130
Title: An Open-label, Phase 0 Clinical Study in Parkinson's Disease Patients and Healthy Volunteers for the Establishment of Biomarker Analytical Methods and ex Vivo Assessment of the Potency of LRRK2 Inhibitors Using Human Biological Samples.
Brief Title: Non-drug Treatment Study in Parkinson's Disease Patients and Healthy Volunteers to Collect Biological Samples in Order to Assess ex Vivo the Activity of Candidate Therapies and Develop Novel Analytical Methods for Biomarkers
Acronym: IRIS-CLE-LRRK2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Servier (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLE-221237-001
Record Dates: First submitted 2023-03-24; First posted 2023-05-01 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Masking Description: Analysis is done ex-vivo and arm assignment is based on if the participant is symptomatic or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Cohort A will include LRRK2 G2019S symptomatic carriers, idiopathic PD patients, and healthy volunteers. It will involve a blood sample collection and an optional cerebrospinal fluid (CSF) collection.
  Interventions: Other: Blood sample collection and an optional cerebrospinal fluid (CSF) collection
- Cohort B (Experimental): Cohort B will include LRRK2 G2019S carriers, idiopathic PD patients, and heathy volunteers. It will involve only a blood sample collection.
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection and an optional cerebrospinal fluid (CSF) collection — No study drug will be administered to study participants.
  Arms: Cohort A
Other: Blood sample collection — No study drug will be administered to study participants.
  Arms: Cohort B

SUMMARY:
This is a non-drug study in patients with Parkinson's Disease (PD) and healthy volunteers to process and analyze their blood and optional cerebrospinal fluid (CSF) samples ex vivo, or outside of their body, to further develop researchers knowledge on LRRK2 biomarkers. Participants were enrolled either in Cohort A or in Cohort B. A blood sample was collected in each participant within a maximum of two study visits within 14 days, and an option to complete both visits on the same day.

DETAILED DESCRIPTION:
This study will allow researchers to assess the potency of investigational LRRK2 inhibitors, outside of participant bodies. It will enroll Parkinson's disease patients (LRRK2 G2019S symptomatic carriers and idiopathic) and healthy volunteers meeting eligibility criteria. The study will consist of a maximum of two study visits, a selection visit to check eligibility criteria, and a sample collection visit. The two visits can take place on the same day or can occur within 14 days of each other. Participants will be assigned to Cohort A or Cohort B, each include a blood sample collection, and an optional cerebrospinal fluid (CSF) collection in Cohort A. No investigational product, study drug, will be administered to study participants.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential (WOCBP) must have a negative pregnancy test
* Parkinson's disease (PD) patients must be at least 40 years old
* Healthy volunteers must be at least 30 years old
* PD patients must have a PD diagnosis, according to the 2015 Movement Disorder Society criteria, with bradykinesia, and at least one of the following: muscular rigidity, or resting tremor with no other suspected cause of Parkinsonism
* The LRRK2 G2019S symptomatic carrier PD patients must have a documented G2019S mutation on the leucine-rich repeat kinase 2 gene (LRRK2)

Exclusion Criteria:

* Pregnant or lactating women
* Have participated in an investigational drug trial within 30 days
* Are SARS-CoV-2, COVID-19, positive within 15 days prior to blood sample collection
* Have another active disease that the investigator believes could interfere with study results

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Assess the potency of LRRK2 inhibitors using target engagement biomarker (cohort B) | Study collection visit Day 1

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalo-Universitaire Grenoble Alpes, La Tronche
  - Centre Hospitalo-Universitaire Lille, Lille
  - Hopital La Pitié Salpétrière-Institut du Cerveau et de la Moelle Epinière-CIC Neurosciences, Paris
  - Centre Hospitalo-Universitaire Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/